CLINICAL TRIAL: NCT06799585
Title: Does Wearing Dental Loupes in Pediatric Dentistry Practice Affect Ergonomic Posture?
Brief Title: Dental Loupes in Pediatric Dentistry Practice Affect Ergonomic Posture
Acronym: ergonomy
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, DİLARA NİL GÜNAÇAR, Assoc. Prof., Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2023/251
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Ergonomics; Musculoskeletal Diseases; Pediatric Dentistry
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- pulpotomy procedures performed with Dental Loupe: Treatment appointments were set to be at the first hour of the day to ensure standardization for each patient. The physicians worked with the same patient chair, physician chair, and DL.
- pulpotomy procedures performed without Dental Loupe: Treatment appointments were set to be at the first hour of the day to ensure standardization for each patient. The physicians worked with the same patient chair, physician chair, without DL.

SUMMARY:
This study aims to investigate the effect of wearing DL on the working posture of pediatric dentists.

DETAILED DESCRIPTION:
In pulpotomy procedures performed with DL in 23 patients and without DL in 23 patients, photographs will taken at a total of 3 times in each patient: at the beginning of the procedure, 15th and 30th minutes. The working postures of the clinicians will analyzed using the Modified-Dental Operator Posture Assessment Instrument (M-DOPAI) method through these photographs.

ELIGIBILITY:
Inclusion Criteria:

* indication for pulpotomy in the mandibular right second primary molar,
* 3 (positive)- 4 (definitely positive) according to the Frankl Behavior Scale,
* parents volunteered to participate in the study and signed the informed consent form,
* did not have any systemic disease or disability.

Exclusion Criteria:

* contraindication for pulpotomy in the mandibular right second primary molar
* 2 (negative)- 1 (definitely negative) according to the Frankl Behavior Scale

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric population
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
The effect of wearing DL on the working posture with Modified-Dental Operator Posture Assessment Instrument (M-DOPAI) | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdoğan University Faculty of Dentistry, Lütfen Seçiniz, Rize Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cinar R, Aydinoglu S, Arslan I, Gunacar DN. Postural effects of dental loupes in pediatric dental practice? BMC Oral Health. 2025 Mar 26;25(1):432. doi: 10.1186/s12903-025-05766-0. PMID 40140822